CLINICAL TRIAL: NCT07221552
Title: Development and Evaluation of PPAL Bedside Commode for Safe Independent Toileting Transfers
Brief Title: Evaluation of the PPAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alicia Koontz (Other)
Collaborators: QUA Inc. (Unknown); National Institute of Nursing Research (NINR) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Alicia Koontz, Professor - School of Health and Rehabilitation Science, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY25100178; 5R44NR019516-03 (NIH)
Record Dates: First submitted 2025-10-24; First posted 2025-10-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Age Problems
Keywords: Activities of daily living; Falls; Assistive technologies

STUDY DESIGN:
Intervention Model Description: This is a single group longitudinal intervention study, conducted using descriptive survey design and data logs by the user.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- PPAL user (Experimental): This is the experimental group. These participants will trial the PPAL.
  Interventions: Device: PPAL

INTERVENTIONS:
Device: PPAL — PPAL is a patented, motorized, height adjustable bedside commode with integrated transfer boards. PPAL incorporates a transfer board that moves up and down as the chair seat is raised or lowered so that the user can always perform a downhill transfer. This innovation will allow individuals with limited mobility who currently rely on caregiver assistance to transfer more independently.

SUMMARY:
This research study is being done to better understand the impact of the PPAL assisted toileting device. The PPAL consists of a powered, height adjustable commode chair with integrated transfer boards. The system is designed to allow the user to assist with their own transfers to/from bed or chair to the PPAL for toileting, with little manual help provided by user's caregivers. Users who require assistance with transfers and their caregivers have a high likelihood of experiencing and injury during transfers.

The purpose of this study is to evaluate the PPAL bedside commode in a home setting to better understand the impact of the device in a 6-week at home trial. Participants will be asked to schedule a home visit with the research team to screen their home and ask questions and observe the participant's current transfer methods to their toilet/commode to ensure that they and the caregiver are an appropriate candidate for the device. Once approved, a delivery date will be arranged to deliver the PPAL to the participant's home. At the end of the 6-week trial, the study team will arrange a final study visit date to retrieve the PPAL and again ask questions and observe a toilet transfer using both the PPAL and the customary commode. Finally, the investigators will interview the participant and the caregiver to ask them about their satisfaction with device. This interview will be audio recorded.

This study involves minimal risks which are expected to occur infrequently. There is the possibility that the participant could obtain a scrape, bruise, cut or pinch injury as you will be working with a device that they are not familiar with. There is also the possibility that the participant could fall when attempting to transfer to or from the device, however the investigators will thoroughly demonstrate the device and monitor your use of it to minimize this risk. There is a risk of breach of confidentiality as text messages and emails may not be encrypted or secure during their transmission or storage and it is possible they could be intercepted and used by others not associated with this study.

There will be no direct benefit to the participant from participating in the study, but it will help the developers of the PPAL better understand the opinions, needs and abilities of the caregivers and patients who may use the device.

ELIGIBILITY:
Toileter Inclusion Criteria:

* Age 18 years or above
* Weighs 300 pounds or less and is able to fit within the dimensions of the PPAL - Has difficulty with getting on or off a toilet or commode at any point in a typical 24-hour period
* Resides in either a home, independent living residence, assisted living or extended care residence
* Able to maintain sitting balance independently (without human assistance) for at least 2 minutes
* If sitting for longer than 2 minutes (with or without assistance), does not get dizzy or lightheaded - residence is able to accommodate the PPAL in the Bedroom or designated space.

Toileter Exclusion Criteria:

* Ventilator users
* Free of acute medical events within the last 3 months
* Had Stage 2 or greater pressure ulcer within the last 3 months
* Upcoming planned medical procedures or surgeries in the next 3 months.

Caregiver Inclusion Criteria:

* Age 18 years or above
* Formal/paid or informal/unpaid caregiver for the patient participant (toileter) who provides toileting assistance at least 3 days per week

Caregiver Exclusion Criteria:

-Physical limitations that prevent caregiver from manually assisting with PPAL transfer or from maneuvering the PPAL around the end-user's residence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in fall efficacy with connection to toileting | Change from pre to post 6 week trial
  We aim to determine whether the use of PPAL reduces fear of falling during toileting activities. To assess this, we will utilize the Fall Concerns Scale for individuals who use Wheelchairs and Scooters (FCS-WC/S). Items are scored on a scale of concern, with 1 being "Not at all concerned" and 4 being "Very Concerned". Scores can be analyzed from specific questions, or the questionnaire as a whole. For this result we will focus on the item specifically associated with getting on/off of a toilet or commode at home. A decrease in FCS-WC/S scores at the end of the study would indicate a reduction in fear of falling.

SECONDARY OUTCOMES:
Change in GG Self-Care score for Toilet Transfer | Change from pre to post 6 week trial
  We aim to observe a change in the GG Self-Care score for toilet transfers, specifically an improvement in the individual's ability to safely get on and off a toilet or commode. This item is scored on a scale from 1 (Dependent: completely reliant on a caregiver) to 6 (Independent: no assistance required). An increase in this score would indicate improved functional independence.
System Usability Scale (SUS) | At the end of the 6 week trial
  We aim to find that PPAL will have at minimum an acceptable level of usability at the end of the trial. The SUS consists of items rated on a scale of 1 (strongly disagree) to 5 (strongly agree), assessing the participants perceived usability of the system in several domain areas. A total score is computed and a score of 68 or higher would be indicative of acceptable usability (scores ranging from 0 to 100 with higher scores indicating better usability).

CONTACTS AND LOCATIONS:
Overall Officials: Alicia M Koontz, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh: Human Engineering Research Laboratories, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Okoli C, Pawlowski SD. The Delphi method as a research tool: an example, design considerations and applications. Information & management. 2004;42(1):15-29.
- [Background] Brown BB. Delphi process: a methodology used for the elicitation of opinions of experts. Rand Corp Santa Monica CA; 1968.
- [Background] Moreland B, Kakara R, Henry A. Trends in Nonfatal Falls and Fall-Related Injuries Among Adults Aged >/=65 Years - United States, 2012-2018. MMWR Morb Mortal Wkly Rep. 2020 Jul 10;69(27):875-881. doi: 10.15585/mmwr.mm6927a5. PMID 32644982
- [Background] Rice L, Kalron A, Berkowitz SH, Backus D, Sosnoff JJ. Fall prevalence in people with multiple sclerosis who use wheelchairs and scooters. Medicine (Baltimore). 2017 Sep;96(35):e7860. doi: 10.1097/MD.0000000000007860. PMID 28858096
- [Background] Kulich HR, Bass SR, Koontz AM. Rehabilitation professional and user evaluation of an integrated push-pull lever drive system for wheelchair mobility. Assist Technol. 2024 Sep;36(5):329-337. doi: 10.1080/10400435.2020.1836068. Epub 2020 Nov 12. PMID 33079646
- [Background] Kulich HR, Bass SR, Griscavage JS, Vijayvargiya A, Slowik JS, Koontz AM. An ergonomic comparison of three different patient transport chairs in a simulated hospital environment. Appl Ergon. 2020 Oct;88:103172. doi: 10.1016/j.apergo.2020.103172. Epub 2020 Jun 8. PMID 32678780
- [Background] Macefield R. How to specify the participant group size for usability studies: a practitioner's guide. Journal of Usability Studies. 2009;5(1):34-45.
- [Background] Demers L, Weiss-Lambrou R, Ska B. The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0): An overview and recent progress. Technology and Disability. 2002;14:101-5.
- [Background] Mortenson WB, Demers L, Fuhrer MJ, Jutai JW, Lenker J, DeRuyter F. Development and preliminary evaluation of the caregiver assistive technology outcome measure. J Rehabil Med. 2015 May;47(5):412-8. doi: 10.2340/16501977-1952. PMID 25783142
- [Background] Boswell-Ruys CL, Harvey LA, Delbaere K, Lord SR. A Falls Concern Scale for people with spinal cord injury (SCI-FCS). Spinal Cord. 2010 Sep;48(9):704-9. doi: 10.1038/sc.2010.1. Epub 2010 Feb 2. PMID 20125107
- [Background] Hittle DF, Shaughnessy PW, Crisler KS, Powell MC, Richard AA, Conway KS, Stearns PM, Engle K. A Study of Reliability and Burden of Home Health Assessment Using OASIS. Home Health Care Serv Q. 2004 Feb 2;22(4):43-63. doi: 10.1300/J027v22n04_03. PMID 29016255
- [Background] Shew PA, Sanders SL, Arthur NC, Bush KW. OASIS inter-rater reliability and reimbursement: a study of inter-rater reliability of the Outcome and Assessment Information Set (OASIS): its effects on the Home Health Resource Group (HHRG) and reimbursement. Home Healthc Nurse. 2010 Jan;28(1):31-6. doi: 10.1097/01.NHH.0000366795.71528.ac. PMID 20032729
- [Background] Sundaram SA, Chung CS, Gebrosky B, Brown J, Grindle GG, Deepak N, Cooper R, Cooper RA. Participatory action design and engineering of a manual wheelchair virtual coach including in-home and community usage. J Spinal Cord Med. 2023 Jul;46(4):546-559. doi: 10.1080/10790268.2022.2107352. Epub 2022 Aug 22. PMID 35994022
- [Background] Daveler B, Gebrosky B, Eckstein I, Cooper R, Grindle GG, Cooper RA. Air-powered shopping carts in grocery stores: a pilot study. Disabil Rehabil Assist Technol. 2022 Jan;17(1):116-122. doi: 10.1080/17483107.2020.1767221. Epub 2020 May 19. PMID 32427527
- [Background] Daveler B, Wang H, Gebrosky B, Grindle GG, Schneider U, Cooper RA. Integration of Pneumatic Technology in Powered Mobility Devices. Top Spinal Cord Inj Rehabil. 2017 Spring;23(2):120-130. doi: 10.1310/sci2302-120. PMID 29339888
- [Background] Grindle GG, Wang H, Jeannis H, Teodorski E, Cooper RA. Design and user evaluation of a wheelchair mounted robotic assisted transfer device. Biomed Res Int. 2015;2015:198476. doi: 10.1155/2015/198476. Epub 2015 Feb 22. PMID 25793190
- [Background] Virzi RA. Refining the Test Phase of Usability Evaluation: How Many Subjects Is Enough? Human Factors. 1992;34(4):457-68.
- [Background] Gagnon MP, Orruno E, Asua J, Abdeljelil AB, Emparanza J. Using a modified technology acceptance model to evaluate healthcare professionals' adoption of a new telemonitoring system. Telemed J E Health. 2012 Jan-Feb;18(1):54-9. doi: 10.1089/tmj.2011.0066. Epub 2011 Nov 14. PMID 22082108
- [Background] Friesen EL. Measuring AT Usability with the Modified System Usability Scale (SUS). Stud Health Technol Inform. 2017;242:137-143. PMID 28873790
- [Background] Sauro J. Measuring Usability with the System Usability Scale (SUS) Measuring 2011
- [Background] Hyman WA. A generic fault tree for medical device error. Journal of Clinical Engineering. 2002;27(2):134-40.
- [Background] Taylor B, Henshall C, Kenyon S, Litchfield I, Greenfield S. Can rapid approaches to qualitative analysis deliver timely, valid findings to clinical leaders? A mixed methods study comparing rapid and thematic analysis. BMJ Open. 2018 Oct 8;8(10):e019993. doi: 10.1136/bmjopen-2017-019993. PMID 30297341
- [Background] Gale RC, Wu J, Erhardt T, Bounthavong M, Reardon CM, Damschroder LJ, Midboe AM. Comparison of rapid vs in-depth qualitative analytic methods from a process evaluation of academic detailing in the Veterans Health Administration. Implement Sci. 2019 Feb 1;14(1):11. doi: 10.1186/s13012-019-0853-y. PMID 30709368
- [Background] Huq MS, Fraass BA, Dunscombe PB, Gibbons JP Jr, Ibbott GS, Medin PM, Mundt A, Mutic S, Palta JR, Thomadsen BR, Williamson JF, Yorke ED. A method for evaluating quality assurance needs in radiation therapy. Int J Radiat Oncol Biol Phys. 2008;71(1 Suppl):S170-3. doi: 10.1016/j.ijrobp.2007.06.081. PMID 18406920
- [Background] Gebrosky B, Pearlman J, Cooper R. Comparison of High-Strength Aluminum Ultralight Wheelchairs Using ANSI/RESNA Testing Standards. Top Spinal Cord Inj Rehabil. 2018 Winter;24(1):63-77. doi: 10.1310/sci16-00057. Epub 2017 Nov 20. PMID 29434462
- [Background] Gebrosky B, Pearlman J, Cooper RA, Cooper R, Kelleher A. Evaluation of lightweight wheelchairs using ANSI/RESNA testing standards. J Rehabil Res Dev. 2013;50(10):1373-89. doi: 10.1682/JRRD.2012.08.0155. PMID 24699973
- [Background] Steinfeld E, Maisel J, Feathers D, D'Souza C. Anthropometry and standards for wheeled mobility: an international comparison. Assist Technol. 2010 Spring;22(1):51-67. doi: 10.1080/10400430903520280. PMID 20402047
- [Background] Noble NL, Sweeney NL. Barriers to the Use of Assistive Devices in Patient Handling. Workplace Health Saf. 2018 Jan;66(1):41-48. doi: 10.1177/2165079917697216. Epub 2017 May 9. PMID 28486032
- [Background] Dicianno BE, Joseph J, Eckstein S, Zigler CK, Quinby EJ, Schmeler MR, Schein RM, Pearlman J, Cooper RA. The future of the provision process for mobility assistive technology: a survey of providers. Disabil Rehabil Assist Technol. 2019 May;14(4):338-345. doi: 10.1080/17483107.2018.1448470. Epub 2018 Mar 20. PMID 29557196
- [Background] Tang K, Diaz J, Lui O, Proulx L, Galle E, Packham T. Do active assist transfer devices improve transfer safety for patients and caregivers in hospital and community settings? A scoping review. Disabil Rehabil Assist Technol. 2020 Aug;15(6):614-624. doi: 10.1080/17483107.2019.1604822. Epub 2019 Jun 28. PMID 31248300
- [Background] Greenhalgh M, Landis JM, Brown J, Kulich H, Bass S, Alqahtani S, Deepak N, Cryzter TM, Grindle GG, Koontz AM, Cooper RA. Assessment of Usability and Task Load Demand Using a Robot-Assisted Transfer Device Compared With a Hoyer Advance for Dependent Wheelchair Transfers. Am J Phys Med Rehabil. 2019 Aug;98(8):729-734. doi: 10.1097/PHM.0000000000001176. PMID 31318755
- [Background] Cohen MH, FAIA F, Nelson GG, Green DA, Borden CM. Patient handling and movement assessments: a white paper. Dallas, TX: The Facility Guidelines Institute. 2010:1-144.
- [Background] Darragh AR, Sommerich CM, Lavender SA, Tanner KJ, Vogel K, Campo M. Musculoskeletal Discomfort, Physical Demand, and Caregiving Activities in Informal Caregivers. J Appl Gerontol. 2015 Sep;34(6):734-60. doi: 10.1177/0733464813496464. Epub 2013 Sep 9. PMID 24652897
- [Background] Owen B, Garg A. Assistive devices for use with patient handling tasks. Advances in Industrial Ergonomics and Safety. 1990;2:585-92.
- [Background] Charney W, Hudson A. Back injury among healthcare workers: Causes, solutions, and impacts: CRC Press; 2003
- [Background] Joey NCM, Ho Marc WK. Does self-initiated sit-to-stand training with an assistive device regain the independence of sit-to-stand in stroke patient? A single-blinded randomized controlled trial. J Rehabil Assist Technol Eng. 2020 Jan 20;7:2055668319866053. doi: 10.1177/2055668319866053. eCollection 2020 Jan-Dec. PMID 32010452
- [Background] Koontz AM, Bass SR, Kulich HR. Accessibility facilitators and barriers affecting independent wheelchair transfers in the community. Disabil Rehabil Assist Technol. 2021 Oct;16(7):741-748. doi: 10.1080/17483107.2019.1710771. Epub 2020 Jan 8. PMID 31913066
- [Background] Toro ML, Koontz AM, Cooper RA. The impact of transfer setup on the performance of independent wheelchair transfers. Hum Factors. 2013 Jun;55(3):567-80. doi: 10.1177/0018720812460549. PMID 23829031
- [Background] Nelson AL, Groer S, Palacios P, Mitchell D, Sabharwal S, Kirby RL, Gavin-Dreschnack D, Powell-Cope G. Wheelchair-related falls in veterans with spinal cord injury residing in the community: a prospective cohort study. Arch Phys Med Rehabil. 2010 Aug;91(8):1166-73. doi: 10.1016/j.apmr.2010.05.008. PMID 20684896
- [Background] Peterson EW, Cho CC, Finlayson ML. Fear of falling and associated activity curtailment among middle aged and older adults with multiple sclerosis. Mult Scler. 2007 Nov;13(9):1168-75. doi: 10.1177/1352458507079260. Epub 2007 Sep 19. PMID 17881391
- [Background] Gavin-Dreschnack D, Nelson A, Fitzgerald S, Harrow J, Sanchez-Anguiano A, Ahmed S, Powell-Cope G. Wheelchair-related falls: current evidence and directions for improved quality care. J Nurs Care Qual. 2005 Apr-Jun;20(2):119-27. doi: 10.1097/00001786-200504000-00006. PMID 15839290
- [Background] Rice L, Kalron A, Berkowitz SH, Backus D, Sosnoff JJ. Fall prevalence in wheeled mobility device users living with multiple sclerosis. Archives of Physical Medicine and Rehabilitation. 2016;97(10):e40-e1.
- [Background] Gagnon D, Koontz A, Mulroy S, Nawoczenski D, Butler-Forslund E, Granstrom A, et al. Biomechanics of sitting pivot transfers among individuals with a spinal cord injury: a review of the current knowledge. Topics in Spinal Cord Injury Rehabilitation. 2009;15(2):33-58.
- [Background] King EC, Holliday PJ, Andrews GJ. Care Challenges in the Bathroom: The Views of Professional Care Providers Working in Clients' Homes. J Appl Gerontol. 2018 Apr;37(4):493-515. doi: 10.1177/0733464816649278. Epub 2016 May 29. PMID 27241041
- [Background] Tzeng HM. A feasibility study of providing folding commode chairs in patient bathrooms to reduce toileting-related falls in an adult acute medical-surgical unit. J Nurs Care Qual. 2011 Jan-Mar;26(1):61-8. doi: 10.1097/NCQ.0b013e3181d94f4d. PMID 22914667
- [Background] Lam K, Shi Y, Boscardin J, Covinsky KE. Unmet Need for Equipment to Help With Bathing and Toileting Among Older US Adults. JAMA Intern Med. 2021 May 1;181(5):662-670. doi: 10.1001/jamainternmed.2021.0204. PMID 33749707
- [Background] Nelson A, Lloyd JD, Menzel N, Gross C. Preventing nursing back injuries: redesigning patient handling tasks. AAOHN J. 2003 Mar;51(3):126-34. PMID 12670100
- [Background] De-Rosende-Celeiro I, Torres G, Seoane-Bouzas M, Avila A. Exploring the use of assistive products to promote functional independence in self-care activities in the bathroom. PLoS One. 2019 Apr 8;14(4):e0215002. doi: 10.1371/journal.pone.0215002. eCollection 2019. PMID 30958846
- [Background] Barrick AL, Rader J, Hoeffer B, Sloane PD, Biddle S. Bathing without a battle: Person-directed care of individuals with dementia: Springer Publishing Company; 2008.
- [Background] Health care workers compensation barometer actuarial analysis. 2018.
- [Background] Garg A, Owen BD, Carlson B. An ergonomic evaluation of nursing assistants' job in a nursing home. Ergonomics. 1992 Sep;35(9):979-95. doi: 10.1080/00140139208967377. PMID 1387079
- [Background] Tsai CY, Boninger ML, Bass SR, Koontz AM. Upper-limb biomechanical analysis of wheelchair transfer techniques in two toilet configurations. Clin Biomech (Bristol). 2018 Jun;55:79-85. doi: 10.1016/j.clinbiomech.2018.04.008. Epub 2018 Apr 12. PMID 29698853
- [Background] Centers for Disease Control and Prevention (CDC). Nonfatal bathroom injuries among persons aged >/=15 years--United States, 2008. MMWR Morb Mortal Wkly Rep. 2011 Jun 10;60(22):729-33. PMID 21659980
- [Background] Sung J, Trace Y, Peterson EW, Sosnoff JJ, Rice LA. Falls among full-time wheelchair users with spinal cord injury and multiple sclerosis: a comparison of characteristics of fallers and circumstances of falls. Disabil Rehabil. 2019 Feb;41(4):389-395. doi: 10.1080/09638288.2017.1393111. Epub 2017 Oct 25. PMID 29069956
- [Background] Blanchet R, Edwards N. A need to improve the assessment of environmental hazards for falls on stairs and in bathrooms: results of a scoping review. BMC Geriatr. 2018 Nov 9;18(1):272. doi: 10.1186/s12877-018-0958-1. PMID 30413144